CLINICAL TRIAL: NCT04267692
Title: Development and Evaluation of Harm Reduction Talking Circles for Urban American Indians and Alaska Natives With Alcohol Use Disorders - Phase III Randomized Clinical Trial
Brief Title: Harm Reduction Talking Circles for American Indians and Alaska Natives With Alcohol Use Disorders
Acronym: HaRTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington State University (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Lonnie Nelson, Associate Professor, Washington State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P60AA026112-RP2; P60AA026112 (NIH)
Record Dates: First submitted 2019-12-16; First posted 2020-02-13 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder
Keywords: Indigenous Medicine; American Indian; Alaska Native; alcohol use disorder; alcohol treatment; treatment efficacy; quality of life; cultural connectedness
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Harm Reduction Treatment Circles (HaRTC) (Experimental): Participants will attend 8, weekly Harm Reduction Treatment Circles. We will not limit participants' access to other treatment or services.
  Interventions: Other: HaRTC

INTERVENTIONS:
Other: HaRTC — HaRT-C participants will attend 8, virtual, adapted, low-barrier, weekly, closed-group Talking Circles-- named Harm Reduction Treatment Circles or HaRTC -- lasting approximately 2 hours each. During the HaRTC, the circle keeper will present the day's harm reduction topic, smudge the space, and allow participants to open themselves up to the circle. Topics presented by the Circle Keeper focus on harm-reduction and improving overall quality of health. Abstinence from alcohol use is not a requirement. We will not limit participants' access to treatment or services in either arm.

SUMMARY:
This randomized clinical trial will compare participants who receive HaRTC versus the nontreatment control arm to see if HaRTC helps urban American Indians and Alaska Natives who meet criteria for an alcohol use disorder to increase their engagement in cultural practices, enhance their quality of life, and reduce their alcohol-related harm.

DETAILED DESCRIPTION:
HaRTC refers to an alcohol treatment that integrates the traditional Native practice of Talking Circles with harm reduction, a low-barrier approach to substance-use treatment that does not require sobriety or use reduction. The HaRTC study is a collaboration between WSU, UW, and Seattle Indian Health Board (SIHB). It is funded by the National Institute on Alcohol Abuse and Alcoholism at the National Institutes of Health. In this study, researchers from WSU and UW are working together with urban-dwelling community members who have Native heritage and lived experience of alcohol use disorder as well as with traditional health professionals, staff and management at SIHB. As a team, we are tailoring, implementing, and evaluating HaRTC as a culturally appropriate treatment for urban American Indians and Alaska Natives.

This study is divided into three phases:

Phase 1: During one-on-one interviews and focus groups, WSU and UW researchers asked patients, traditional healers, staff and management at SIHB how to best tailor HaRTC.

Phase 2: The researchers assembled a community action board comprised of Native community members who have lived experience as well as traditional health professionals, staff and management at SIHB to refine the HaRTC treatment manual and procedures to best fit the needs, setting and values at SIHB based on their own lived experiences and on the findings from Phase 1. This protocol was then revisited together with our community action board and community partners to ensure appropriate physical distancing in the wake of the COVID-19 pandemic. Thus, our in-person procedures were converted to a fully virtual, online protocol.

Phase 3: Researchers are conducting a randomized clinical trial of the virtual adapted Harm Reduction Treatment Circles (HaRTC) program. Participants (N=280) in the RCT will be urban American Indians and Alaska Natives. Additionally, they must be at least 21 years of age and meet criteria for a current alcohol use disorder. Participants will provide informed consent and will be randomized (like flipping a coin) to receive either HaRTC or no-treatment control so the investigators can evaluate whether HaRTC is efficacious. Participants will be asked questions about their involvement in cultural practices, alcohol use and quality of life prior to randomization, a month into the HaRTC, after the HaRTC ends, and at 1-, 3-, and 6-month follow-up interviews. It is expected that HaRTC will help patients increase their engagement with cultural traditions, enhance their quality of life, and reduce their experience of alcohol-related harm. If so, the research team will work with SIHB to make this intervention sustainable for its community members.

ELIGIBILITY:
Inclusion Criteria:

1. being urban AI/AN,
2. being at least 21 years of age (for legal reasons), and
3. meeting criteria for a current AUD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)

Exclusion Criteria:

1. refusal or inability to consent to participation in research, and
2. potential to place the safety or security of other patients or staff at risk

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol frequency | Pre-intervention, mid-, immediate post-intervention, 1 month post-intervention, 3 months post intervention, and 6 months post-intervention.
  Alcohol and Substance Use Frequency Assessment items were adapted from the Addiction Severity Index-Fifth Edition (ASI-5th Ed) and will be used to assess frequency of alcohol use in the past 30 days. Scores range from 0 to 30 with higher scores indicating more frequent drinking.
Change in Peak alcohol use | Pre-intervention, mid-, immediate post-intervention, 1 month post-intervention, 3 months post intervention, and 6 months post-intervention.
  The Alcohol Quantity and Use Assessment was created by the research team for previous studies with a similar population and will be used to record the quantity of alcohol consumed on participants' heaviest, typical, and lightest drinking days in the past month. Scores are expressed in number of standard drinks with higher numbers indicating heavier drinking.
Change in Alcohol-related harm | Pre-intervention, mid-, immediate post-intervention, 1 month post-intervention, 3 months post intervention, and 6 months post-intervention.
  The Short Inventory of Problems-2nd Revision (SIP-2R), a psychometrically reliable and valid 15-item, Likert-scale questionnaire, measures social, occupational, and psychological problems related to alcohol use. Scores range from 0 to 45 with higher scores indicating more severe alcohol-related harm.
Change in EuroQoL-5 Dimensional-5 Level | Pre-intervention, mid-, immediately post-intervention, 1 month post-intervention, 3 months post intervention, and 6 months post-intervention.
  The EuroQoL-5 Dimensional-5 Level is a widely used generic measure of health status consisting of two parts. The first part (the descriptive system) assesses health in five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT, ANXIETY / DEPRESSION), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). Each domain is rated on a 5 point likert scale. Scores range from 5-25, with higher scores indicating poorer health related quality of life.
Change in Cost effectiveness | 6 months before study participation compared to 6 months after enrollment.
  **Self-report data for cost-effectiveness analyses
  -The Non-Study Resources Form: documents change in medical and nonmedical resources used by participants.
Change in Ethyl glucuronide | Pre-intervention, mid-, immediately post-intervention, 1 month post-intervention, 3 months post intervention, and 6 months post-intervention.
  Ethyl glucuronide (EtG) urine tests will be used to validate self-reported alcohol use at each assessment. EtG, a metabolite of ethyl alcohol formed in the body after ethanol exposure, reflects alcohol consumption over the previous 72 hours. EtG (cutoff 300 mg/nl) will serve as a secondary outcome in analyses.

OTHER OUTCOMES:
Change in Cultural connectedness | Pre-intervention, mid-, immediately post-intervention, 1 month post-intervention, 3 months post intervention, and 6 months post-intervention.
  The Cultural Connectedness Scale is a 29-item Likert type measure consisting of 3 dimensions: identity, traditions, and spirituality. Scores can range from 29-145, with higher scores indicating a greater degree of cultural connectedness. Criterion validity was demonstrated with cultural connectedness dimensions adequately correlating with other indicators of wellness. The resulting scale scores will represent the proposed mediator in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie A Nelson, PhD, Principal Investigator — Washington State University
Locations (1):
- Seattle Indian Health Board, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
According to the data MOU signed by the 3 collaborating institutions, SIHB owns the data and grants researchers at WSU and UW the right to maintain a copy of data to use up to 6 years following study completion to fulfill study aims. Thereafter, SIHB will maintain sole ownership of and access to the data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT04267692/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT04267692/ICF_000.pdf